CLINICAL TRIAL: NCT04806854
Title: A Single-Center, Randomized, Open-Label, Parallel Arm Study of Daily Oral LUM-201 in Naive-to-Treatment, Prepubertal Children With Idiopathic Pediatric Growth Hormone Deficiency (PGHD)
Brief Title: PK and PD Study of LUM-201 in Children With Idiopathic Growth Hormone Deficiency: (OraGrowtH212)
Acronym: OraGrowtH212
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lumos Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUM-201-03
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Growth Hormone Deficiency
Keywords: GHD, PGHD, LUM-201, growth hormone secretagogue, height, catch-up growth, pulsatility, pharmacokinetics, pharmacodynamics, PK, PD, idiopathic
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LUM-201 (1.6 mg/kg/day) (Experimental)
  Interventions: Drug: LUM-201
- LUM-201 (3.2 mg/kg/day) (Experimental)
  Interventions: Drug: LUM-201

INTERVENTIONS:
Drug: LUM-201 — Administered orally once daily

SUMMARY:
The goals of this single site trial are to study the pharmacokinetics (PK) and pharmacodynamics of LUM-201 and effects of LUM-201 administration on growth hormone release over time in children with idiopathic pediatric growth hormone deficiency (PGHD).

DETAILED DESCRIPTION:
This trial will have a single screening visit to assess if subjects are eligible to start study therapy. Once subjects have completed screening, and if they are determined to be eligible, they will return to the clinic for a 12-hour pulsatility study. On Day Two of the trial, subjects will be randomized to receive one of two oral daily doses of LUM-201 and PK samples will be collected. All subjects will have an equal chance of being placed in either of the two groups.

The trial consists of treatment until subjects achieve near adult height. After screening, subjects will return to the clinic monthly for the first 6 visits and every three months thereafter. At most clinic visits, subjects will have a physical exam, blood and urine collections. At the Month 6 visit subjects will repeat the 12-hour pulsatility and PK studies.

ELIGIBILITY:
Inclusion Criteria:

* Have a chronological age ≥ 4.0 years and ≤ 10.0 years for girls and ≤ 12.0 years for boys.
* Have a minimum body weight of 16 kg at the time of screening.
* Have a bone age examination at screening or within the 6 months prior to screening that is delayed with respect to chronological age. Bone age should be based on the apparent BA of the proximal and distal phalanges, as opposed to the metacarpals, carpals and distal forearm. A central BA reader will make the final determination on BA eligibility.
* Have HT-SDS ≤ -2.0 or a HT-SDS ≥ 2 SD below mean parental HT-SDS. If the other data (slow HV, low IGF-1, peak GH < 10, and 6-month BA delay) are all consistent with idiopathic GHD, the subject may be enrolled with a height SDS > -2.0 after consultation with the MMs.
* Have an accurate baseline height velocity ≤ 5.5 cm/year based on at least 6-months of growth, if available
* Within the past 6 months have a maximal GH response > 3 and < 10 ng/mL from at least one prior GH stimulation test within the past 6 months
* Have prepubertal status as evidenced by Tanner Stage I breast development in girls and testicular volume < 4.0 mL in boys.
* Have an arm span to height ratio > 96.5%
* In girls, have genetic testing results to rule out Turner syndrome. If SHOX genetic testing results are available, they need to be negative.
* Have normal thyroid function. Subjects diagnosed with hypothyroidism must have documented successful treatment for at least 30 days prior to the Baseline visit.

Exclusion Criteria:

* Any medical or genetic condition which, in the opinion of the PI or Medical Monitor (MM), can be an independent cause of short stature and/or limit the response to exogenous growth factor treatment (e.g., diabetes, , idiopathic short stature (ISS), SHOX-deficiency, skeletal dysplasia, constitutional growth delay, SGA, other).
* A medical or genetic condition that, in the opinion of the PI and/or MM, adds unwarranted risk to use of LUM-201 (e.g., scoliosis).
* Use of any medication that, in the opinion of the PI and/or MM, can independently cause short stature or limit the response to exogenous growth factors (e.g., glucocorticoids).
* Evidence or history of an intracranial mass (e.g., pituitary tumor, craniopharyngioma).
* Prior treatment with growth factors including, but not limited to, GH, IGF-1, and GH secretagogues. (These may be used for limited times as a diagnostic test.)
* Suspicion of absence of pituitary function as evidenced by a maximal stimulated GH ≤ 3 ng/mL or pituitary hormone deficiencies beyond GH and thyroid function or a diagnosis of Organic PGHD.
* At birth, gestational age < 36.0 weeks.
* Participation in any therapeutic trial of investigational drug(s) within the prior 6 months.
* History of spinal, cranial or total body irradiation.
* Recent commencement of non-stimulant therapy to treat attention deficit hyperactivity disorder (ADHD).

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Augmented Growth Hormone (GH) Pulsatility | Day 1 to Month 6
  12-hour mean GH concentration
Pharmacokinetics of LUM-201 and M8 | Day 1 to Month 6
  Plasma concentrations (Cmax/Steady State)

SECONDARY OUTCOMES:
Incidence of adverse events in children with idiopathic GHD | up to 8 years
  Number of events
Height standard deviation score (SDS) | Day 1 to Month 12
  Change in HT-SDS from Baseline to Month 6 and Month 12

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Maternal and Child Research, University of Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No